CLINICAL TRIAL: NCT01423500
Title: Allogeneic Stem Cell Transplantation in Children and Adolescents With Acute Lymphoblastic Leukaemia
Brief Title: ALL-SCT BFM International- HSCT in Children and Adolescents With ALL
Acronym: ALL-SCT-BFMi
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: St. Anna Kinderkrebsforschung (Other)
Responsible Party: Principal Investigator, Prof. Christina Peters, MD, PhD, Children's Cancer Research Institute, Austria
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EudraCT 2005-005106-23
Record Dates: First submitted 2011-08-23; First posted 2011-08-26 (Estimated); Last update posted 2015-06-26 (Estimated); Status verified 2015-06

CONDITIONS: Lymphoblastic Leukemia, Acute, Childhood;
Keywords: ALL; HSCT; children; adolescents
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Etoposide; Whole-Body Irradiation; fludarabine; Muromonab-CD3; treosulfan; Thiotepa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- MSD - Matched Sibling Donor (Other): patients with a MSD receive a conditioning of TBI (12 Gy, 6 fractions) and VP16 60mg/kg for one day (-3)
  Interventions: Drug: VP16; Radiation: TBI
- MD - Matched Donor (Other): patients with a HLA matched unrelated Donor (9/10 oder 10/10) receive TBI (12Gy in 6 fractions), VP16 60mg/kg/d on day -3 and ATG fresenius 20mg/kg/d on day -3,-2,-1
  Interventions: Drug: VP16, ATG; Radiation: TBI
- MMD - Mismatched Donor (Other): Patients with a MMD receive stem cells either from cord blood, a haploidentical donor (parent) or from a non-related donor with a match less or equal 8/10
  Interventions: Drug: Fludarabine, OKT3, Treosulfan, Thiotepa; Drug: VP16, ATG; Radiation: TBI

INTERVENTIONS:
Drug: VP16 — patients with MSD receive as conditioning VP16 60mg/kg/d on day -3
  Other Names: Etoposid
  Arms: MSD - Matched Sibling Donor
Radiation: TBI — patients with a MSD receive TBI (12Gy in 6 fractions) as conditioning
  Other Names: Total body irradiation
  Arms: MSD - Matched Sibling Donor
Drug: VP16, ATG — patients with a HLA matched unrelated Donor (9/10 oder 10/10) receive VP16 60mg/kg/d on day -3 and ATG fresenius 20mg/kg/d on day -3,-2,-1
  Other Names: Etoposid, Antithymoglobuline
  Arms: MD - Matched Donor
Radiation: TBI — patients with a HLA matched unrelated Donor (9/10 oder 10/10) receive TBI (12Gy in 6 fractions)
  Other Names: total body irradiation
  Arms: MD - Matched Donor
Drug: Fludarabine, OKT3, Treosulfan, Thiotepa — patients with a MMD (haploidentical or cord blood) receive Fludarabine 30mg/m²/d on day -9 to -5, ATG fresenius 20mg/kg/d on day -3,-2,-1, Treosulfan 14g/m²/d on day -7 to -5 and Thiotepa 2x5mg/kg/d on day -4
  Other Names: ATG: Antithymoglobuline
  Arms: MMD - Mismatched Donor
Drug: VP16, ATG — patients with MMD-transplantation (8/10)receive VP16 60mg/kg/d on day -4, ATG from day -3 to day-1 20mg/kg/d
  Other Names: VP16: Etoposid; ATG: Antithymoglobuline
  Arms: MMD - Mismatched Donor
Radiation: TBI — patients with a MMD-transplantation (8/10) receive 12 Gy in 6 fractions
  Other Names: TBI: total body irradiation
  Arms: MMD - Mismatched Donor

SUMMARY:
With this protocol the ALL-SCT BFM international study group wants

* to evaluate whether hematopoietic stem cell transplantation (HSCT) from matched family or unrelated donors (MD) is equivalent to the HSCT from matched sibling donors (MSD).
* to evaluate the efficacy of hematopoietic stem cell transplantation (HSCT)from mismatched family or unrelated donors (MMD) as compared to HSCT from matched sibling donors or matched donors.
* to determine whether therapy has been carried out according to the main HSCT protocol recommendations. The standardisation of the treatment options during HSCT from different donor types aims at the achievement of an optimal comparison of survival after HSCT with survival after chemotherapy only.
* to prospectively evaluate and compare the incidence of acute and chronic Graft-versus-Host-Disease (GvHD) after HSCT from matched sibling donor (MSD), from matched donor (MD) and from mismatched donor (MMD).

DETAILED DESCRIPTION:
Patients with high risk or relapsed acute lymphoblastic leukaemia (ALL) have a worse prognosis compared to all other patients with ALL. For these patients additional therapy approaches are required after they have achieved remission with multimodal chemotherapy. Allogeneic haematopoetic stem cell transplantation shows promising results mainly due to an immunological antileukaemic control by the graft-versus-leukaemia effect but treatment related mortality and morbidity remains a serious problem.

ELIGIBILITY:
Inclusion Criteria:

* age at time of initial diagnosis or relapse diagnosis, respectively under or equal 18 years
* indication for allogeneic hematopoietic stem cell transplantation(HSCT)
* complete remission before hematopoietic stem cell transplantation (HSCT)
* written consent of the parents (legal guardian) and, if necessary, the minor patient via Informed Consent Form
* no pregnancy
* no secondary malignancy
* no previous hematopoietic stem cell transplantation (HSCT)
* hematopoietic stem cell transplantation (HSCT) is performed in a study participating centre.

Exclusion Criteria:

* age at time of initial diagnosis or relapse diagnosis, respectively above 18 years
* no indication for allogeneic HSCT
* no complete remission before SCT
* no written consent of the parents (legal guardian) and, if necessary, the minor patient via Informed Consent Form
* pregnancy
* secondary malignancy
* previous HSCT
* HSCT is not performed in a study participating centre.

Ages: 3 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 405 (Estimated)
Dates: Start 2007-01; Primary Completion 2011-09 (Actual); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Event free survival | 10 years
  Event-free and overall survival after allogeneic HSCT

SECONDARY OUTCOMES:
number of patients with GvHD acute and chronic Graft-versus-Host-Disease (GvHD) | 10 years
  evaluation of the incidence and severity of acute Grade I-IV graft versus Host disease and of limited or extensive chronic graft versus host disease
occurrence and course of late effects after chemotherapy with subsequent allogeneic HSCT | 10 years
  evaluation of organ dysfunctions according to WHO Toxicity score
occurrence and course of late effects after chemotherapy with subsequent allogeneic HSCT | 10 years
  evaluation of growth retardation and endocrine dysfunction
occurrence and course of late effects after chemotherapy with subsequent allogeneic HSCT | 10 years
  Evaluation of incidence of aseptic bone necrosis.
occurrence and course of subsequent malignancies after chemotherapy with subsequent allogeneic HSCT | 10 years
  Evaluation of incidence of secondary cancer after total body irradiation and/or chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Christina Peters Peters, Prof MD PHD, Study Chair — St. Anna Kinderkrebsforschung; Petr Sedlacek, Prof. MD, Principal Investigator — Department of Paediatric Haematology and Oncology. HSCT Unit Prague; Marianne Ifversen, MD, Principal Investigator — Paediatric Clinic II, Rigshospitalet Copenhagen; Jean-Hugues Dalle, Prof. MD, Principal Investigator — HSCT Unit Robert Debré Hospital Paris; Jerry Stein, Prof. MD, Principal Investigator — Schneider Children's Medical Center, Israel; Adriana Balduzzi, MD, Principal Investigator — Ospedale San Gerardo Monza; Marc Bierings, MD, Principal Investigator — Wilhelmina Children's Hospital Utrecht; Jacek Wachowiak, MD, Prof., Principal Investigator — Department of Paediatric Oncology, Haematology and Transplantology, University of Medical Sciences Poznan; Sabina Sufliarska, MD, Principal Investigator — HSCT Unit, University Children's Hospital Bratislava; Jacek Toporski, MD, Principal Investigator — Department of Paediatric Oncology Lund; Sema Anak, Prof MD, Principal Investigator — Paediatric HSCT Unit, Istanbul School of Medicine; Akif Yesilipek, MD Prof, Principal Investigator — Dep. of Paediatric Haematology-Oncology and HSCT, Akdeniz University School of Medicine
Locations (24):
- Austria (3):
  - Universitätsklinik für Kinder- und Jugendheilkunde, Klin. Abt. f. Hämato-Onkologie, Graz
  - Universitätsklinik für Kinder- und Jugendheilkunde, Innsbruck
  - St. Anna Children's Hospital, Vienna
- Department of Paediatric Haematology and Oncology HSCT-Unit, Prague, Czechia
- Pediatric Clinic II, Rigshospitalet, Copenhagen, Denmark
- Pediatric Immuno-Hematology Unit Robert Debré Hospital, Paris, France
- Israel (2):
  - Rambam Medical Center, Haifa
  - Schneider Children's Medical Center of Israel, Petah Tikva
- Clinica Pediatrica dell'Universita di Milano Bicocca, Hospitale San Gerardo, Monza, Italy
- Netherlands (3):
  - Leiden University Hospital, Leiden
  - Radboud University - Nijmegen Medical Centre, Nijmegen
  - Department of Paediatric Haematology and Oncology, Wilhelmina Children's Hospital, Utrecht
- Poland (5):
  - University Hospital, Collegium Medicum UMK, Pediatric Hematology and Oncology, Bydgoszcz
  - Department of Transplantation, University Children's Hospital, Krakow
  - Children's University Hospital - Hematology - Oncology, Lublin
  - Department of Pediadric Oncology, Hematology and Transplantology, University of Medical Sciences, Poznan
  - Wroclaw Medical University, Dept. of Children Hematology and Oncology, Wroclaw
- Department of Pediatric Bone Marrow Transplantation Unit, University Childrens´ Hospital, Bratislava, Slovakia
- Department of Pediatric Oncology, Lund University Hospital, Lund, Sweden
- Turkey (Türkiye) (5):
  - Department of Pediatrics, Gülhane Military Medical Academy, Ankara
  - Dept. of Paediatrics - BMT Unit, School of Medicine, University of Ankara, Ankara
  - Department of Pediatric Hematology-Oncology and Pediatric Stem Cell Transplantation, Akdeniz University School of Medicine, Antalya
  - Department of Pediatric Hematology, Oncology and BMT, Istanbul School of Medicine, Istanbul
  - Pediatric BMT Centre, Ege University, Izmir

REFERENCES:
- [Result] Peters C, Schrauder A, Schrappe M, von Stackelberg A, Stary J, Yaniv I, Gadner H, Klingebiel T; BFM Study Group, the IBFM-Study Group and the Paediatric Disease Working Party of the EBMT. Allogeneic haematopoietic stem cell transplantation in children with acute lymphoblastic leukaemia: the BFM/IBFM/EBMT concepts. Bone Marrow Transplant. 2005 Mar;35 Suppl 1:S9-11. doi: 10.1038/sj.bmt.1704835. PMID 15812540
- [Result] Pulsipher MA, Peters C, Pui CH. High-risk pediatric acute lymphoblastic leukemia: to transplant or not to transplant? Biol Blood Marrow Transplant. 2011 Jan;17(1 Suppl):S137-48. doi: 10.1016/j.bbmt.2010.10.005. PMID 21195303
- [Result] Peters C, Schrappe M, von Stackelberg A, Schrauder A, Bader P, Ebell W, Lang P, Sykora KW, Schrum J, Kremens B, Ehlert K, Albert MH, Meisel R, Matthes-Martin S, Gungor T, Holter W, Strahm B, Gruhn B, Schulz A, Woessmann W, Poetschger U, Zimmermann M, Klingebiel T. Stem-cell transplantation in children with acute lymphoblastic leukemia: A prospective international multicenter trial comparing sibling donors with matched unrelated donors-The ALL-SCT-BFM-2003 trial. J Clin Oncol. 2015 Apr 10;33(11):1265-74. doi: 10.1200/JCO.2014.58.9747. Epub 2015 Mar 9. PMID 25753432
- [Derived] Tasian SK, Peters C. Targeted therapy or transplantation for paediatric ABL-class Ph-like acute lymphocytic leukaemia? Lancet Haematol. 2020 Dec;7(12):e858-e859. doi: 10.1016/S2352-3026(20)30369-0. No abstract available. PMID 33242441
- [Derived] Balduzzi A, Dalle JH, Wachowiak J, Yaniv I, Yesilipek A, Sedlacek P, Bierings M, Ifversen M, Sufliarska S, Kalwak K, Lankester A, Toporski J, Di Maio L, Glogova E, Poetschger U, Peters C. Transplantation in Children and Adolescents with Acute Lymphoblastic Leukemia from a Matched Donor versus an HLA-Identical Sibling: Is the Outcome Comparable? Results from the International BFM ALL SCT 2007 Study. Biol Blood Marrow Transplant. 2019 Nov;25(11):2197-2210. doi: 10.1016/j.bbmt.2019.07.011. Epub 2019 Jul 15. PMID 31319153